CLINICAL TRIAL: NCT06941844
Title: A Phase 3 Multicenter, Randomized, Double-blind, Placebo-controlled, 12-Week Study (Part A) With a 40-Week Open-label Extension (Part B) Evaluating the Efficacy and Safety of Oral MM120 Compared to Placebo in the Treatment of Adults With Major Depressive Disorder - Emerge
Brief Title: A Phase 3 Trial of MM120 for Major Depressive Disorder (Emerge)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Definium Therapeutics US, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MM120-310
Record Dates: First submitted 2025-04-16; First posted 2025-04-24 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-05

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 - Placebo (Placebo Comparator): A substance that is designed to have no therapeutic value
  Interventions: Other: Placebo
- Arm 2 - 100µg MM120 (LSD D-Tartrate) (Experimental): A psychoactive substance that mediates effects mainly through an agonist activity in the serotonin 2A receptor (5-HT2A)
  Interventions: Drug: MM120 (LSD D-Tartrate)

INTERVENTIONS:
Other: Placebo — A substance that is designed to have no therapeutic value
  Arms: Arm 1 - Placebo
Drug: MM120 (LSD D-Tartrate) — A psychoactive substance that mediates effects mainly through an agonist activity in the serotonin 2A receptor (5-HT2A)
  Arms: Arm 2 - 100µg MM120 (LSD D-Tartrate)

SUMMARY:
A Phase 3 Double-blind, Placebo-controlled Study (Part A) with an Open-label Extension (Part B) Evaluating MM120 Compared to Placebo in Major Depressive Disorder - Emerge

DETAILED DESCRIPTION:
The study will enroll approximately 140 adult men and women aged 18 to 74 years, inclusive with a Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) confirmed primary diagnosis of MDD,a minimum MADRS total score of at least 26 and a CGI-S score of at least 4 at Screening and Baseline without clinically relevant medical or psychiatric history.

The study consists of a 12-week randomized, double-blind, single-dose administration period evaluating MM120 versus placebo, followed by a 40-week extension phase with the opportunity for open-label treatment. During this phase, participants will be monitored and evaluated for potential treatment with MM120 based on pre-specified safety and symptom severity criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of MDD per DSM-5
2. Male or female aged 18 to 74
3. Currently experiencing a major depressive episode (MDE) of ≥8 weeks and ≤24 months duration
4. MADRS Total Score ≥26
5. CGI-S Score ≥4

Exclusion Criteria:

1. Certain psychiatric disorders (other than major depressive disorder)
2. First degree relative with or lifetime history of a psychotic disorder or bipolar disorder
3. Current diagnosis of alcohol or substance use disorder (excluding nicotine and caffeine
4. Any clinically significant unstable illness

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Montgomery-Åsberg Depression Rating Scale (MADRS) total score at Week 6 | Baseline to Week 6
  The MADRS is used to assess depression severity and to detect changes due to antidepressant treatment. The MADRS includes 10 clinician-completed items. Each of the 10 questions is scored with a range of 0-6 points. An item score of 0 indicates item not present or normal, while an item score of 6 indicates severe or continuous presence of the symptoms. The total possible score is 60, and higher scores represent a more severe condition.

SECONDARY OUTCOMES:
Change from Baseline in the MADRS total score at Week 12, Week 4, Week 2, and Week 1 | Week 12, Week 4, Week 2, and Week 1
  The MADRS is used to assess depression severity and to detect changes due to antidepressant treatment. The MADRS includes 10 clinician-completed items. Each of the 10 questions is scored with a range of 0-6 points. An item score of 0 indicates item not present or normal, while an item score of 6 indicates severe or continuous presence of the symptoms. The total possible score is 60, and higher scores represent a more severe condition.
MADRS response (reduction from Baseline score of ≥50%) at each timepoint assessed during the 12-week double-blind period | Baseline to Week 12
  The MADRS is used to assess depression severity and to detect changes due to antidepressant treatment. The MADRS includes 10 clinician-completed items. Each of the 10 questions is scored with a range of 0-6 points. An item score of 0 indicates item not present or normal, while an item score of 6 indicates severe or continuous presence of the symptoms. The total possible score is 60, and higher scores represent a more severe condition.
MADRS remission (total score ≤10) at each timepoint assessed during the 12-week double-blind treatment period | Baseline to Week 12
  The MADRS is used to assess depression severity and to detect changes due to antidepressant treatment. The MADRS includes 10 clinician-completed items. Each of the 10 questions is scored with a range of 0-6 points. An item score of 0 indicates item not present or normal, while an item score of 6 indicates severe or continuous presence of the symptoms. The total possible score is 60, and higher scores represent a more severe condition.
Clinical Global Impression - Improvement (CGI-I) Scale score at each timepoint assessed during the 12-week double-blind period | Day 2 to Week 12
  The CGI-I scale is used to measure the clinician's assessment of how much the participant's illness has improved or worsened relative to Baseline (Visit 2). The CGI-I comprises one item with 7 possible ratings (1-7 points), where a lower score indicates improvement, and a higher score indicates worsening.
Change from Baseline throughout the 12-week double-blind period at each timepoint assessed in Clinical Global Impression - Severity (CGI-S) Scale score | Baseline to Week 12
  The CGI-S scale assesses the clinician's impression of the participant's current severity of illness relative to the clinician's experience with patients who have the same diagnosis. The CGI-S comprises one item with 7 possible ratings (1-7 points), where a higher score indicates more severe illness.
Change from Baseline throughout the 12-week double-blind period at each timepoint assessed in Patient Global Impression - Severity (PGI-S) Scale score | Baseline to Week 12
  The PGI scale is the patient-reported outcome (PRO) counterpart to the CGI scale. The PGI-S comprises one participant-completed item with 5 possible ratings (1-5) where a higher score indicates more severe illness.
Change from Baseline throughout the 12-week double-blind period at each timepoint assessed in MADRS-6 | Baseline to Week 12
  The MADRS-6 is a subscale of the 10-item MADRS and evaluates the core symptoms of depression: apparent sadness, reported sadness, inner tension, lassitude, inability to feel, and pessimistic thought.
Change from Baseline throughout the 12-week double-blind period at each timepoint assessed in Hamilton Anxiety Rating Scale (HAM-A) | Baseline to Week 12
  The HAM-A consists of the following 14 items that encompass both psychological and somatic symptoms of anxiety. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Change from Baseline throughout the 12-week double-blind period at each timepoint assessed in -Work Productivity and Activity Impairment Questionnaire (WPAI) | Baseline to Week 12
  The WPAI-SHP is a 6-item questionnaire, with a recall period of the past 7 days. The WPAI measures impairments in both paid work and unpaid work. It measures absenteeism, presenteeism as well as impairment in unpaid activity because of the health problem under study.
Change from Baseline throughout the 12-week double-blind period at each timepoint assessed in -EuroQol-5 Dimensions - 5 Levels (EQ-5D-5L) | Baseline to Week 12
  The EuroQol 5 Dimension 5 Level (EQ-5D-5L) is a self-reported outcome measure used to evaluate health outcomes over a wide range of health conditions and treatments. The EQ-5D consists of the EQ-5D descriptive system and the EQ visual analogue scale (VAS).
Change from Baseline in the Changes in Sexual Functioning Questionnaire (CSFQ-14) total score at each timepoint assessed during the double-blind period | Baseline to Week 12
  The CSFQ-14 is a structured self-reported questionnaire designed to measure illness- and medication-related changes in sexual functioning that consists of 14 items measuring sexual functioning as a total score (14 items). There is a male and female version of the CSFQ-14 scale and a total score of less than 47 for men and less than 41 for women indicates sexual dysfunction. Lower scores are associated with worsened sexual functioning.
Percent of men and women with normal and abnormal sexual functioning at each timepoint assessed during the double-blind period | Baseline to Week 12
  The CSFQ-14 is a structured self-reported questionnaire designed to measure illness- and medication-related changes in sexual functioning that consists of 14 items measuring sexual functioning as a total score (14 items). There is a male and female version of the CSFQ-14 scale and a total score of less than 47 for men and less than 41 for women indicates sexual dysfunction. Lower scores are associated with worsened sexual functioning.
Percent of participants requiring one, two, three, four, or five doses of MM120 during the 52-week study (Part A and Part B) as assessed by participants meeting protocol-specified retreatment criteria during the 40-week open-label period | Day 1 to Week 52
  Percent of participants requiring one, two, three, four, or five doses of MM120 during the 52-week study (Part A and Part B) as assessed by participants meeting protocol-specified retreatment criteria during the 40-week open-label period.
Time to first treatment or lack of efficacy in the open-label period (Part B) | Day 1 to Week 52
  Measured as time from first dosing in the Double-blind period to participant meeting MADRS criteria for re-dose or meeting criteria for lack of efficacy.
Need for MM120 treatment as assessed by the average number of MM120 treatments during the study | Day 1 to Week 52
  Average number of treatments assessed from first dose in the double-blind period through completion of the open label extension.
MADRS response (reduction from Baseline score of ≥50%) at each timepoint assessed during the 40-week open-label period | 40-week open label period
  The MADRS is used to assess depression severity and to detect changes due to antidepressant treatment. The MADRS includes 10 clinician-completed items. Each of the 10 questions is scored with a range of 0-6 points. An item score of 0 indicates item not present or normal, while an item score of 6 indicates severe or continuous presence of the symptoms. The total possible score is 60, and higher scores represent a more severe condition.
MADRS remission (total score ≤10) at each timepoint assessed during the 40-week open-label period | 40-week open label period
  The MADRS is used to assess depression severity and to detect changes due to antidepressant treatment. The MADRS includes 10 clinician-completed items. Each of the 10 questions is scored with a range of 0-6 points. An item score
Change from Double-blind Baseline throughout the 40-week open-label period at each timepoint assessed in MADRS total score | Baseline to Week 52
  The MADRS is used to assess depression severity and to detect changes due to antidepressant treatment. The MADRS includes 10 clinician-completed items. Each of the 10 questions is scored with a range of 0-6 points. An item score of 0 indicates item not present or normal, while an item score of 6 indicates severe or continuous presence of the symptoms. The total possible score is 60, and higher scores represent a more severe condition.
Change from Double-blind Baseline throughout the 40-week open-label period at each timepoint assessed in Clinical Global Impression - Severity (CGI-S) Scale score | Baseline to Week 52
  The CGI-S scale assesses the clinician's impression of the participant's current severity of illness relative to the clinician's experience with patients who have the same diagnosis. The CGI-S comprises one item with 7 possible ratings (1-7 points), where a higher score indicates more severe illness.
Change from Double-blind Baseline throughout the 40-week open-label period at each timepoint assessed in Patient Global Impression - Severity (PGI-S) Scale score | Baseline to Week 52
  The PGI scale is the patient-reported outcome (PRO) counterpart to the CGI scale. The PGI-S comprises one participant-completed item with 5 possible ratings (1-5) where a higher score indicates more severe illness.
Change from Double-blind Baseline throughout the 40-week open-label period at each timepoint assessed in MADRS-6 total score | Baseline to Week 52
  The MADRS-6 is a subscale of the 10-item MADRS and evaluates the core symptoms of depression: apparent sadness, reported sadness, inner tension, lassitude, inability to feel, and pessimistic thought.
Change from Double-blind Baseline throughout the 40-week open-label period at each timepoint assessed in HAM-A total score | Baseline to Week 52
  The HAM-A consists of the following 14 items that encompass both psychological and somatic symptoms of anxiety. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Change from Double-blind Baseline throughout the 40-week open-label period at each timepoint assessed in WPAI | Baseline to Week 52
  The WPAI-SHP is a 6-item questionnaire, with a recall period of the past 7 days. The WPAI measures impairments in both paid work and unpaid work. It measures absenteeism, presenteeism as well as impairment in unpaid activity because of the health problem under study.
Change from Double-blind Baseline throughout the 40-week open-label period at each timepoint assessed in EQ-5D-5L | Baseline to Week 52
  The EuroQol 5 Dimension 5 Level (EQ-5D-5L) is a self-reported outcome measure used to evaluate health outcomes over a wide range of health conditions and treatments. The EQ-5D consists of the EQ-5D descriptive system and the EQ visual analogue scale (VAS).
CSFQ-14 total score at each timepoint assessed during the open-label period | 40 week open label period
  The CSFQ-14 is a structured self-reported questionnaire designed to measure illness- and medication-related changes in sexual functioning that consists of 14 items measuring sexual functioning as a total score (14 items). There is a male and female version of the CSFQ-14 scale and a total score of less than 47 for men and less than 41 for women indicates sexual dysfunction. Lower scores are associated with worsened sexual functioning.
Percent men and women with normal and abnormal sexual functioning at each timepoint assessed during the open-label period | 40 week open label period
  The CSFQ-14 is a structured self-reported questionnaire designed to measure illness- and medication-related changes in sexual functioning that consists of 14 items measuring sexual functioning as a total score (14 items). There is a male and female version of the CSFQ-14 scale and a total score of less than 47 for men and less than 41 for women indicates sexual dysfunction. Lower scores are associated with worsened sexual functioning.

CONTACTS AND LOCATIONS:
Locations (28):
- United States (28):
  - Preferred Research Partner, Fayetteville, Arkansas
  - Preferred Research Partners, Inc, Little Rock, Arkansas
  - Kadima Neuropsychiatry Institute, La Jolla, California
  - Psychedelic Science Institute, Santa Monica, California
  - Mountain View Clinical Research, Inc, Denver, Colorado
  - Clinical Neuroscience Solutions, Inc, Jacksonville, Florida
  - Segal Trials- Center for Psychedelic Research, Lauderhill, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - Charter Research, Orlando, Florida
  - Uptown Research, Chicago, Illinois
  - Sheppard Pratt, Baltimore, Maryland
  - Adams Clinical Boston, Boston, Massachusetts
  - Adams Clinical, Watertown, Massachusetts
  - University of Missouri, Columbia, Missouri
  - Cenexel HRI, Berlin, New Jersey
  - Spectrum Neuroscience and Treatment Institute, New York, New York
  - Adams Clinical Harlem, New York, New York
  - Columbia - New York State Psychiatric Institute, New York, New York
  - Neuro-Behavioral Clinical Research, Canton, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Adams Clinical Philadelphia, Philadelphia, Pennsylvania
  - Scranton Medical Institute, LLC, Scranton, Pennsylvania
  - Clinical Neuroscience Solutions, Inc, Memphis, Tennessee
  - Dell Medical School, University of Texas at Austin, Austin, Texas
  - Austin Clinical Trial Partners, Austin, Texas
  - FutureSearch Trials of Dallas, Dallas, Texas
  - Cedar Clinical Research, Murray, Utah
  - Memory Clinic, Inc, Bennington, Vermont